CLINICAL TRIAL: NCT03453632
Title: Evaluation of the Efficacy of Injections of Botulinic Toxin in Plantar Lesions of Patients Suffering From Localized Epidermolysis Bullosa Simplex : Double Blind Randomized Controlled Study.
Brief Title: Injections of Botulinic Toxin in Plantar Lesions of Localized Epidermolysis Bullosa Simplex
Acronym: EBTox
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RC31/16/8917; 2017-002332-16 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-03-05 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Epidermolysis Bullosa Simplex
Keywords: Dermatology; Rare skin diseases; epidermolysis bullosa simplex; botulinic toxin; blisters
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Blister | interventions — abobotulinumtoxinA; Drugs, Investigational

STUDY DESIGN:
Intervention Model Description: Each subject is his own witness, receiving the 2 treatments : left foot vs. right foot
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinic toxin (Experimental): Injections of botulinic toxin (Dysport®, Allergan) 200 UI
  Interventions: Drug: Botulinic toxin
- Placebo (Placebo Comparator): Injections of physiological serum
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinic toxin — Clinical photographs of the soles Standardized anesthesia protocol (lidocaine, prilocaine on soles, cryo-spray, oral administration of paracetamol and only if necessary oxycodone and hydroxyzine).
  Cleaning and antiseptic on the soles Injections of botulinic toxin (200 UI) on right or left foot
  Other Names: Dysport® (experimental drug)
  Arms: Botulinic toxin
Drug: Placebo — Clinical photographs of the soles Standardized anesthesia protocol (lidocaine, prilocaine on soles, cryo-spray, oral administration of paracetamol and only if necessary oxycodone and hydroxyzine).
  Cleaning and antiseptic on the soles Injections of physiological serum (200 UI) on right or left foot
  Other Names: physiological serum
  Arms: Placebo

SUMMARY:
The investigators hypothesize that palmar injections of botulinic toxin, via an inhibition of the sudation, would limit the occurrence of blisters in localized epidermolysis bullosa simplex (LEBS).

DETAILED DESCRIPTION:
Epidermolysis bullosa is a group of rare genetic diseases characterized by the occurrence of blisters and erosions due to skin fragility. There are 4 different subgroups, based on the location of the skin cleavage area. The most frequent subgroup is the simplex form, consisting predominantly of the localized form (localized epidermolysis bullosa simplex: LEBS). The incidence of LEBS was estimated at between 1/318.000 and 1/35.000. The disease starts early in infancy by the occurrence of blisters and erosions located on soles, secondary to frictions during the walk. The phenomenon is worsened by heat and sudation. LEBS is due to mutations in keratin genes. Life expectancy in LEBS is normal but the quality of life is significantly impaired due to permanent skin pain and limitation of everyday activities (walking, sports). There is no effective or curative treatment. Patients must limit the frictions, protect the skin and use plasters in case of skin lesions.

Botulinic toxin has an agreement for the treatment of axillary hyperhidrosis and has been shown to be also effective on palms and soles. The efficacy of botulinic toxin in plantar lesions of LEBS has been reported in the literature (one case report and a short retrospective series of 6 patients) but there is no proper study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LEBS based on clinical symptoms and in some cases histological or molecular findings
* Palmar skin lesions: blisters and/or : erosions, edematous and erythematous lesions, crusts. 3 lesions per foot, as a minimum
* Similar clinical severity of skin lesions on both feet
* Patient with social security
* Written consent of the patient
* Patient able to understand the study's questionnaires

Exclusion Criteria:

* Patients with only one leg and a different number of toes on each foot.
* Known hypersensitivity to botulinic toxin or its excipients
* Current treatment with aminosides
* Myasthenia
* Swallowing difficulties
* Respiratory disorders
* Past medical history of dysphagia or pneumopathy of inhalation
* Known allergy or contraindications to lidocaine, prilocaine, paracetamol or nitrous oxide
* Pregnancy (positive pregnancy test (β-HCG) for women of childbearing age, performed within the 2 days prior to the study. Breastfeeding.
* Contraception during 6 months from inclusion
* Mental or physical or judicial incapacity to fill the questionnaires
* Guardianship patients
* Skin infection on the soles at the time of the inclusion
* Skin lesions located on the soles, not related to LEBS (ie. post traumatic wound, wart)
* Patient suffering from dishydrosis
* Botulinic toxin injections in the previous 6 months
* Inclusion in another study in the previous 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Global clinical improvement on each foot assessed by a blinded centralized independent reviewer using photographs, at M3 vs.baseline: IGA score (Improvement Global Assessment) assessed for each foot | at baseline vs month 3
  IGA score is a 5-point scale (range from 0 to 4): 0=no improvement or worsening / 1=minimal improvement / 2=moderate improvement / 3=significant improvement / 4=total disappearance

SECONDARY OUTCOMES:
Global clinical improvement on each foot assessed by a blinded centralized independent reviewer using photographs: IGA score (Improvement Global Assessment) for each foot | at baseline vs month 6
  IGA score is a 5-point scale (range from 0 to 4): 0=no improvement or worsening / 1=minimal improvement / 2=moderate improvement / 3=significant improvement / 4=total disappearance
Global clinical improvement on each foot assessed by the investigator: IGA score (Improvement Global Assessment) assessed for each foot. | at month1, month 3 and month 6 respectively vs baseline
  IGA score is a 5-point scale (range from 0 to 4): 0=no improvement or worsening / 1=minimal improvement / 2=moderate improvement / 3=significant improvement / 4=total disappearance
Efficacy assessment concerning the number of plantar lesions clinically observed by the investigator | at baseline, month 1, month 3 and month 6
  on each foot (erythematous and edematous areas, blisters, skin erosion, crusts)
Efficacy assessment on each foot of the affected plantar skin surface (blisters, erosions, erythematous and edematous areas, crusts) | at baseline, month 1, month 3 and month 6
  calculation of this affected surface by delimiting its contours on a standardized photography using "Image J" software = computerized assessment by a blinded centralized independent reviewer.
Efficacy assessment by the patient himself, for each foot | at month 1, month 3, month 6 and month 9
  Global improvement assessed with a 5-point score (0=no improvement or worsening / 1=minimal improvement / 2=moderate improvement / 3=significant improvement / 4=total disappearance)
Plantar pain assessment by the patient himself, for each foot | at baseline, month 1, month 3 and month 6
  Plantar pain assessment , using a 0 to 10 pain EVA scale. To perform the assessment, patient is requested to be standing on one foot (assessment of pain felt for this foot using EVA scale) then, standing on the other foot (assessment of pain felt for this other foot using EVA scale).
Immediate tolerance during injection : | Day 0
  Assessment performed by the patient of the pain felt during the act for each foot, using a 0 to 10 pain EVA scale (patient interview). Assessment performed by the investigator of local adverse events (for each foot) or general adverse events, during the injections
Mid-term and long-term tolerance | Day 0, month 1, month 3 and month 6 and month 9
  Assessment performed by the patient of local adverse events (for each foot) or general adverse events reported in the home patient's diary between the protocol visits (collected at month 1, month 3, month 6 and month 9). • Assessment performed by investigator of local adverse events (for each foot) or general adverse events, at D0 (at the end of/after the injections), M3 and M6.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Mazereeuw-Hautier, MD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - University Hospital Bordeaux, Bordeaux
  - University Hospital Nice, Nice
  - Saint-Louis Hospital - APHP, Paris
  - Hôpital Larrey - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fine JD, Bruckner-Tuderman L, Eady RA, Bauer EA, Bauer JW, Has C, Heagerty A, Hintner H, Hovnanian A, Jonkman MF, Leigh I, Marinkovich MP, Martinez AE, McGrath JA, Mellerio JE, Moss C, Murrell DF, Shimizu H, Uitto J, Woodley D, Zambruno G. Inherited epidermolysis bullosa: updated recommendations on diagnosis and classification. J Am Acad Dermatol. 2014 Jun;70(6):1103-26. doi: 10.1016/j.jaad.2014.01.903. Epub 2014 Mar 29. PMID 24690439
- [Background] Sprecher E. Epidermolysis bullosa simplex. Dermatol Clin. 2010 Jan;28(1):23-32. doi: 10.1016/j.det.2009.10.003. PMID 19945613
- [Background] Langan SM, Williams HC. A systematic review of randomized controlled trials of treatments for inherited forms of epidermolysis bullosa. Clin Exp Dermatol. 2009 Jan;34(1):20-5. doi: 10.1111/j.1365-2230.2008.02789.x. Epub 2008 Sep 25. PMID 18828848
- [Background] Abitbol RJ, Zhou LH. Treatment of epidermolysis bullosa simplex, Weber-Cockayne type, with botulinum toxin type A. Arch Dermatol. 2009 Jan;145(1):13-5. doi: 10.1001/archdermatol.2008.546. No abstract available. PMID 19153338
- [Background] Schwieger-Briel A, Chakkittakandiyil A, Lara-Corrales I, Aujla N, Lane AT, Lucky AW, Bruckner AL, Pope E. Instrument for scoring clinical outcome of research for epidermolysis bullosa: a consensus-generated clinical research tool. Pediatr Dermatol. 2015 Jan-Feb;32(1):41-52. doi: 10.1111/pde.12317. Epub 2014 Mar 20. PMID 24650374